CLINICAL TRIAL: NCT04133610
Title: HPVPro Study: Comparison of HPV Detection in Clinician-collected Cervical Swabs and Self-sampled Cervicovaginal Swabs
Acronym: HPVPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: National Institute for Cancer Research, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 343
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Cervical Cancer; Cervical Dysplasia; Human Papillomavirus Infection
Keywords: human papillomavirus; HPV; self-sampling; cervical swab; cervicovaginal swab; cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-sampling device in media (Experimental): Women will undergo clinician-obtained cervical swab and self-sampled cervicovaginal swab using self-sampling device in STM media. HPV will be detected by hybridization technique.
  Interventions: Diagnostic Test: Self-sampling using digene HC2 DNA Collection Device
- Dry self-sampling device (Experimental): Women will undergo clinician-obtained cervical swab and self-sampled cervicovaginal swab using dry self-sampling device. HPV will be detected by hybridization and PCR techniques.
  Interventions: Diagnostic Test: Self-sampling using Evalyn Brush

INTERVENTIONS:
Diagnostic Test: Self-sampling using digene HC2 DNA Collection Device — All women will undergo a clinician-collected cervical swab and self-collected cervicovaginal swab.
  Arms: Self-sampling device in media
Diagnostic Test: Self-sampling using Evalyn Brush — All women will undergo a clinician-collected cervical swab and self-collected cervicovaginal swab.
  Arms: Dry self-sampling device

SUMMARY:
Comparison of the detection of human papillomavirus DNA in paired physician-obtained cervical swabs and self-sampled cervicovaginal swabs and evaluation of HPV prevalence in Czech women screening population.

DETAILED DESCRIPTION:
The cervical screening program in the Czech Republic is based on cytology with HPV triage. Nevertheless, cytology-based cervical screening may switch to HPV-based cervical screening in future. The implementation of primary HPV screening and insuficiency cervical screening attendance are a major challenge. The offering of self-sampling to the cervical screening non-attenders could increase women's participation as was shown in several European countries. The objective of the HPVPro study was to find out the HPV prevalence in the screening population of Czech women since there are no data for the Czech Republic. The second objective was to compare HPV DNA detection rate in paired self-sampled cervicovaginal swabs and physician-obtained cervical swabs and to determine acceptability of self-sampling HPV DNA test by Czech women. This information is important for optimisation of cervical cancer screening program in the Czech Republic.

ELIGIBILITY:
Inclusion Criteria:

* Women with age 30-64 years.
* Women attending cervical cancer screening program in Czech Republic.
* Women with completed informed consent.

Exclusion Criteria:

* Pregnant women.
* Women with no sexual intercourse experience.
* Women after cervical conization or hysterectomy.
* Women with CIN or cervical carcinoma in anamnesis.
* Women at risk of increased bleeding.

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1044 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
HPV prevalence | 18 months
  Evaluation of the prevalence of high-risk human papillomavirus infection in screening population of Czech women.
Concordance of HPV positivity in self-collected cervicovaginal swabs and clinician-collected cervical swabs | 18 months
  Paired cervical and cervicovaginal swabs will be collected in the same day and will be tested by the same method. Concordance of HPV positivity in both swabs will be evaluated.

SECONDARY OUTCOMES:
Comparison of different human papillomavirus DNA detection methods in cervical and cervicovaginal swabs. | 18 months
  Hybridization and PCR-based HPV detection methods will be tested in both cervical and cervicovaginal swabs and results of these two methods will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD, PhD., Study Director — Palacky University in Olomouc, Faculty of Medicine and Dentistry
Locations (3):
- Czechia (3):
  - GYN-PREN, Ltd., Frýdek-Místek
  - GYNPRENATAL, Ltd., Havířov
  - MEDIOL, Ltd., Olomouc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaworek H, Bouska O, Kourilova P, Hajduch M, Koudelakova V. High-risk HPV prevalence in the Czech cervical cancer screening population: a comparison of clinician-collected and self-collected sampling. Eur J Public Health. 2025 Aug 1;35(4):760-765. doi: 10.1093/eurpub/ckaf045. PMID 40194781